CLINICAL TRIAL: NCT05219812
Title: A Randomized, Double-blind, Cross-over, Placebo-controlled, Multi-center, Phase 2a Study to Assess the Safety and Signal in Efficacy of BAY 2395840 in Patients With Diabetic Neuropathic Pain
Brief Title: A Study to Learn How Safe BAY2395840 is and How Well it Works in Participants Who Have Diabetic Nerve Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19636; 2021-001392-17 (EudraCT Number)
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Neuropathic Pain Associated With Diabetic Peripheral Neuropathy; Peripheral Neuropathic Pain; Diabetes Mellitus
Keywords: Neuropathic Pain
MeSH Terms: conditions — Diabetes Mellitus; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (BAY2395840 - placebo) (Experimental): Participants will be randomly assigned to treatment regimen of double-blind BAY2395840, and after an interim single blind period for washout will switch to double-blind placebo.
  Interventions: Drug: BAY2395840; Drug: Placebo for BAY2395840
- Group 2 (Placebo - BAY2395840) (Experimental): Participants will start with a treatment regimen of double-blind placebo, and after an interim single blind period for washout will switch to double-blind BAY2395840.
  Interventions: Drug: BAY2395840; Drug: Placebo for BAY2395840

INTERVENTIONS:
Drug: BAY2395840 — Tablet, intake orally.
Drug: Placebo for BAY2395840 — Tablet, intake orally.

SUMMARY:
Researchers are looking for a better way to treat people who have diabetic neuropathic pain (DNP), a condition in which diabetes results in pain due to nerve damage.

People with diabetes have high blood sugar levels. Over the time, high blood sugar levels can cause damage to the nerves in the body, which results in DNP. The nerve damage in this condition is localized in a stocking and glove like pattern and starts in the feet and can move upwards on your legs. Some patients also progress having pain in their fingers/hands. People with DNP have pain in these areas as well as reduction/loss of feeling, and at times light touch can feel like pain.

In this study, the researchers want to learn more about a new study treatment called BAY 2395840. BAY 2395840 works by blocking a receptor called the bradykinin B1 receptor, or B1R. This receptor is has been shown to play a role in pain perception.

The researchers also want to learn how well BAY 2395840 helps to reduce pain in the study participants. To answer this question, the researchers will measure how the participants' pain changes after taking BAY 2395840 compared to a placebo. A placebo looks like a treatment but does not have any medicine in it. The researchers also want to learn how safe BAY 2395840 is for the participants to take.

The study will include adults.

This will be a "crossover" study. In a crossover study, all the participants will receive both treatments (BAY 2395840 and placebo), but in a different order. All participants in this study will take BAY 2395840 and a placebo as tablets by mouth.

There will be 2 periods in the study. Participants taking BAY 2395840 during period 1 will switch to placebo during period 2 and vice versa. There will some time for the switch from one period to another to make sure that whatever tablet you received in period 1 is gone from your system before period 2 starts to allow for the best possible evaluation of each tablet without any confusing effects.

The study is double blinded meaning that neither you nor your doctor will know which drug you are on. The sequence of double-blind placebo and BAY treatment will be determined randomly by a computerized system.

During the study, the participants will visit their study site 13 times. Each participant will be in the study for about 16 weeks. The treatment duration will be about 11 weeks.

During the study, the study team will:

* take blood and urine samples
* do physical examinations
* check the participants' overall health
* check the participants' heart health using an electrocardiogram (ECG)
* ask the participants about any medications they have been taking, and what adverse events they are having

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age at the time of signing the informed consent.
* Have documented diagnosis of type 1 OR type 2 diabetes mellitus (DM).
* Have painful distal symmetrical sensorimotor diabetic neuropathy for at least 6 months prior to the screening and confirmed at screening via the modified Toronto Clinical Neuropathy Score with a score of at least 3.
* Weekly mean 24-hour average pain Numeric Rating Scale (NRS) ≥ 4 with adequate variability (not the same score on all daily pain ratings) and compliance (non-missing pain score on at least 6 out of 7 consecutive days) in daily pain recording during the 7-day NRS baseline period.
* Neuropathic pain according to the Douleur Neuropathique 4 Questions (DN4 questionnaire) at screening visit with a score of at least 4 out of 10.
* Participant should be on stable antidiabetic treatment for at least 3 months prior to the screening visit and there should be no pre-planned changes to antidiabetic treatment during this study.
* Participant is willing to use only rescue medication provided by the site and is willing to withdraw temporarily all other neuropathic pain medications which were in use before study participation.
* Participant is willing and able to use the electronic hand-held device on their own.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Clinically significant cardiovascular or cerebrovascular disease including Acute coronary syndrome (ACS)/myocardial infarction /stroke/Transient ischemic attack (TIA) within previous 3 months before screening visit.
* Major depressive episode within 6 months prior to screening. Patients with stable depression and on stable antidepressant dose (no change in medication and /or dosing regimen) for the past 6 months are allowed to participate, provided the antidepressant used is not listed under prohibited medications.
* Any differential diagnosis of peripheral diabetic neuropathy (PDN) including but not limited to other neuropathies (e.g. vitamin B12 deficiency, Chronic Inflammatory Demyelinating Polyneuropathy), polyradiculopathies, central disorders (e.g. demyelinating disease), or rheumatological disease (e.g. foot arthritis, plantar fasciitis).
* Concurrent malignancy or history of cancer (exception of basal cell or squamous cell carcinoma of the skin) within the last 5 years prior to screening.
* Any other diseases or conditions that according to the investigator can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study intervention (e.g. chronic bowel disease, Crohn's disease, and ulcerative colitis).
* Any serious or unstable diseases or conditions including psychiatric disorders that might interfere with the conduct of the study or the interpretation of the results.
* Major surgery or radiological procedures (e.g. Percutaneous transluminal angioplasty (PTA) and stenting of peripheral vascular lesions in lower extremities) within 3 months before screening visit or scheduled during the study period, which might interfere pain response evaluation.
* Symptomatic peripheral arterial disease in lower or upper extremities, including diabetic ulcers.
* Use of live, attenuated, replication-competent vaccines.
* Previous use of strong opioids (e.g. oxymorphone, oxycodone) for neuropathic pain anytime, or topical use of capsaicin within 3 months prior to the screening visit.
* History or current diagnosis of electrocardiogram (ECG) abnormalities indicating significant risk of safety for study participants.
* Moderate-to-severe hepatic impairment defined as Child-Pugh Class B or C.
* Have platelets ≤ 100 x 109/L, or neutrophil count < 1.2 x 109/L (or equivalent), hemoglobin ≤ 100 g/L for women or hemoglobin ≤ 110 g/L for men at screening.
* Glycemic control unstable (hemoglobin HbA1c ≥11% or 97 mmol/mol) within 3 months prior to screening (e.g. ketoacidosis requiring hospitalization, any recent episode of hypoglycemia requiring assistance through medical intervention, uncontrolled hyperglycemia).
* ALT >2xULN, or AST >2xULN, or total bilirubin greater than ULN, or alkaline phosphatase (AP) >2x ULN, or INR greater than ULN (unless related to anticoagulation treatment) at screening.
* Positive hepatitis B virus surface antigen (HBsAg) or positive hepatitis C virus antibodies (anti-HCV) and detection of mRNA (HCV-mRNA tested only if hepatitis C virus antibodies detected).
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2 calculated by Modification of Diet in Renal Disease (MDRD) formula.
* Uncontrolled hypertension despite optimal treatment with antihypertensive(s), indicated by a sitting systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 110 mmHg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Change in weekly mean 24-hour average pain intensity score using the 11-point Numeric Rating Scale (NRS) from baseline to the end of intervention | Baseline to end of intervention (in total up to 16 weeks)
  NRS is an one-item assessment of average neuropathic pain intensity which is presented as an 11-point Likert scale with 0 as "no pain" and 10 as "worst imaginable pain".

SECONDARY OUTCOMES:
Change in Neuropathic Pain Symptom Inventory (NPSI) score from baseline to the end of intervention. | At visit 2, visit 4, visit 6, visit 8, visit 10 and at visit 12 end of intervention (EOI).
  The Neuropathic Pain Symptom Inventory (NPSI) is a PRO developed to evaluate different symptoms of neuropathic pain.
Change in Patient Global Impression of Severity (PGI-S) score from baseline to the end of intervention. | At visit 2, visit 4, visit 6, visit 8, visit 10 and at visit 12 end of intervention (EOI).
  The PGI-S is a one-item self-reported instrument used to assess to assess patients' impression of disease severity with a 6-point scale response options, scores ranging from 1 ("none") to 6 ("very severe).
The proportion of participants achieving a ≥30% and a ≥50% reduction in weekly mean 24-hour average pain intensity score (i.e. responder rates using NRS) | From baseline to end of intervention (in total up to 12 weeks)
Number of participants with treatment emergent adverse events (TEAE) | From start of study intervention to 14 days after last dose.

CONTACTS AND LOCATIONS:
Locations (30):
- Czechia (7):
  - NEUROHK s.r.o, Choceň
  - Interni a diabetologicka ambulance - Krnov, Krnov
  - Fakultni nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Praglandia, Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
  - Diabetologicka ambulance Vlasim, Vlašim
- Germany (6):
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe, Baden-Wurttemberg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover, Lower Saxony
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Herz- und Diabeteszentrum Nordrhein-Westfalen (HDZ NRW), Bad Oeynhausen, North Rhine-Westphalia
  - InnoDiab Forschung GmbH, Essen, North Rhine-Westphalia
  - Klinische Forschung Berlin GbR, Berlin
- Hungary (3):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Clinexpert Kft., Budapest
  - Coromed Smo Kft, Pécs
- Slovakia (6):
  - ALIAN s.r.o., Bardejov
  - NEUROPOINT sro, Neurologicka ambulancia, Bratislava
  - Internal and Diabetes Clinic - IN-DIA s.r.o. | Lucenec, Slovakia, Lučenec
  - Vseobecna nemocnica v Ziari nad Hronom, Žiar nad Hronom
  - Neuron - D.T. sro, Neurologicka ambulancia, Žilina
  - Medivasa s.r.o., Žilina
- Spain (5):
  - Gerencia de Gestion Integrada A Coruna | Department of Endocrinology and Nutrition, A Coruña, A Coruña
  - Complexo HU Ferrol | Endocrinología y Nutrición, Ferrol, A Coruña
  - Hospital Univ. Bellvitge | Anestesiología y Unidad del Dolor, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Gregorio Maranon | Endocrinology Department, Madrid
- United Kingdom (3):
  - MAC Clinical Research - Teesside, Teesside, Stockton-on-Tees
  - King's College Hospital - NHS Foundation Trust, London
  - MAC Research Centre - Manchester, Manchester

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Stemper B, Lowen S, Fritsch A, Hoffmann A, Sarkar A. The bradykinin-1 receptor antagonist fulmetibant in patients with diabetic neuropathic pain: the randomized, crossover, placebo-controlled, double-blind, phase 2a BRADiNP study. Pain. 2025 Oct 1;166(10):2421-2429. doi: 10.1097/j.pain.0000000000003642. Epub 2025 May 6. PMID 40334047
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/19636
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/